CLINICAL TRIAL: NCT00285038
Title: US-Doppler for the Diagnosis of Asymptomatic DVT in Gynecologic Cancer Patients
Brief Title: Ultrasound (US)-Doppler for the Diagnosis of Asymptomatic Deep Vein Thrombosis (DVT) in Gynecologic Cancer Patients
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr Beck-Razi, Rambam Medical Center
Other Study IDs: NIRACTIL
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2006-01

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Gynecological cancer
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The aim of this study is to determine the prevalence of asymptomatic lower extremity DVT detected by Doppler ultrasound in a selected group of patients suffering from gynecological malignancies.

DETAILED DESCRIPTION:
The association between malignancy and venous thromboembolism (VTE) is well known. It has been shown that there is a high prevalence of VTE in gynecological malignancies. Early detection of VTE can identify patients who may benefit from anticoagulant therapy and prevent morbidity and mortality.

NO clear guidelines are available for anticoagulant prophylaxis in a selected group of ambulatory gynecological cancer patients. It has been shown, in other selected groups of patients that Ultrasound Doppler can be used in order to diagnose asymptomatic DVT (deep vein thrombosis).

ELIGIBILITY:
Inclusion Criteria:

* Gynecological cancer patients
* Ambulatory performance status of 0-2
* Prior to, or during, chemotherapy and/or radiation

Exclusion Criteria:

* Before or near surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecological Ambulatory cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nira Beck-Razi, MD, Principal Investigator — Ministry of Health, Israel
Locations (1):
- Rambam Medical Center, Haifa, Israel